CLINICAL TRIAL: NCT00980057
Title: Adaptive Cardiac Resynchronization Therapy Study
Acronym: aCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Adaptive CRT
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adaptive CRT (aCRT) arm (Experimental): Intervention: Cardiac resynchronization therapy (CRT-D) with Adaptive CRT algorithm ON
  Interventions: Device: Adaptive CRT (aCRT)
- Echo-optimized arm (Active Comparator): Intervention: Cardiac resynchronization therapy (CRT-D) with standard biventricular pacing (Adaptive CRT algorithm OFF)
  Interventions: Device: Echo

INTERVENTIONS:
Device: Adaptive CRT (aCRT) — Adaptive CRT (aCRT) is an algorithm, which provides ambulatory adjustment of pacing configuration (LV-only or BiV) and AV and VV delays based on periodic automatic evaluation of electrical conduction to optimize cardiac function
  Other Names: aCRT
  Arms: Adaptive CRT (aCRT) arm
Device: Echo — Standard BiV pacing with settings optimized using a standardized echocardiographic protocol
  Other Names: Control
  Arms: Echo-optimized arm

SUMMARY:
The purpose of this study is to demonstrate the AdaptivCRT algorithm is at least as good as manual echo based optimization in regard to patient outcomes and cardiac performance

DETAILED DESCRIPTION:
The trial has 3 primary end points:

* to demonstrate that over 6-month follow-up, the proportion of the patients improved in the aCRT arm is at least as high as in the Echo arm
* to demonstrate that cardiac function is similar when using aCRT versus echo-optimized settings
* to demonstrate that aCRT does not result in inappropriate AV or VV delay settings

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign and date the study Informed Consent form
* Subject is at least 18 years of age (or older, if required by local law)
* Subject is expected to remain available for at least six months of follow-up visits
* Subject is indicated for a study device that will be implanted within 30 days after signing the Informed Consent form
* Subject has an intrinsic QRS duration greater than or equal to 120 milliseconds (documented within 30 days prior to enrollment)
* Subject has a left ventricular ejection fraction less than or equal to 35 percent (method per physician discretion) (documented within 180 days prior to enrollment)
* Subject is diagnosed with New York Heart Association (NYHA) class III or IV (within 30 days prior to enrollment) despite optimal medical therapy which is defined as: ACE-inhibitor (Angiotensin-Converting Enzyme) or Angiotensin II Receptor Blocker (ARB), if tolerated, for at least one month prior to implant, AND beta-blocker for at least three months preceding implant, if tolerated, and stable for one month, OR subject has an urgent medical need for an implantable cardioverter defibrillator (ICD) that precludes waiting the one or three months for the medication requirements for ACE inhibitor, ARB or beta-blocker

Exclusion Criteria:

* Subject has chronic (permanent) atrial arrhythmias for which pharmacological therapy and/or cardioversion have been unsuccessful or have not been attempted
* Subject has existing CRT system
* Subject has non-intact or unstable leads
* Subject has medical conditions that would limit study participation (per physician discretion)
* Subject is enrolled in one or more concurrent studies that would confound the study results of this study as determined by Medtronic
* Subject has unstable angina, or experienced an acute myocardial infarction (MI) or received coronary artery revascularization (CABG) or coronary angioplasty (PTCA) (documented within 30 days prior to enrollment)
* Subject has a mechanical right heart valve or is scheduled to undergo valve repair or valve replacement during the course of the study
* Subject is post-heart transplant (subjects on the heart transplant list for the first time are not excluded)
* Subject has a limited life expectancy that would not allow completion of the 6 month visit
* Subject is pregnant (In the United States, all women of child-bearing potential must undergo a pregnancy test within seven days prior to aCRT download into device)
* Subject meets the exclusion criteria required by local law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2011-08-04 (Actual); Study Completion 2012-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adaptive CRT Trial Leader, Study Chair — Medtronic
Locations (105):
- United States (55):
  - Huntsville, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Glendale, California
  - San Bernardino, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Clearwater, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Augusta, Georgia
  - Barrington, Illinois
  - Fort Wayne, Indiana
  - Davenport, Iowa
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Takoma Park, Maryland
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Saginaw, Michigan
  - Saint Cloud, Minnesota
  - Saint Louis Park, Minnesota
  - Saint Paul, Minnesota
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Morristown, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - New York, New York
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Charleston, South Carolina
  - Spartanburg, South Carolina
  - Chattanooga, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Tyler, Texas
  - Burlington, Vermont
  - Norfolk, Virginia
  - Richmond, Virginia
  - Bellingham, Washington
  - Spokane, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Australia (6):
  - Adelaide
  - Camperdown
  - Chermside
  - Darlinghurst
  - Perth
  - Spring Hill
- Linz, Austria
- Belgium (3):
  - Genk
  - Leuven
  - Yvoir
- Canada (6):
  - Calgary
  - London
  - Montreal
  - Newmarket
  - Ottawa
  - Victoria
- Denmark (4):
  - Aalborg
  - Aarhus
  - Copenhagen
  - Odense
- Germany (5):
  - Bochum
  - Hamburg
  - Lüdenscheid
  - Reinbek
  - Trier
- Athens, Greece
- Hong Kong, Hong Kong
- Budapest, Hungary
- Italy (4):
  - Milan
  - Pavia
  - Pedara
  - Rozzano
- Japan (3):
  - Osaka
  - Tokyo
  - Tsukuba
- Netherlands (2):
  - Nijmegen
  - Rotterdam
- Norway (2):
  - Bergen
  - Oslo
- Tyumen, Russia
- Riyadh, Saudi Arabia
- Serbia (3):
  - Belgrade
  - Kamenitz
  - Niš
- Spain (4):
  - Albacete
  - Madrid
  - Majadahonda
  - Vitoria-Gasteiz
- Sweden (2):
  - Lund
  - Stockholm

REFERENCES:
- [Derived] Gasparini M, Birnie D, Lemke B, Aonuma K, Lee KL, Gorcsan J 3rd, Landolina M, Klepfer R, Meloni S, Cicconelli M, Grammatico A, Martin DO. Adaptive Cardiac Resynchronization Therapy Reduces Atrial Fibrillation Incidence in Heart Failure Patients With Prolonged AV Conduction: The Adaptive CRT Randomized Trial. Circ Arrhythm Electrophysiol. 2019 May;12(5):e007260. doi: 10.1161/CIRCEP.119.007260. No abstract available. PMID 30991823
- [Derived] Birnie D, Hudnall H, Lemke B, Aonuma K, Lee KL, Gasparini M, Gorcsan J 3rd, Cerkvenik J, Martin DO. Continuous optimization of cardiac resynchronization therapy reduces atrial fibrillation in heart failure patients: Results of the Adaptive Cardiac Resynchronization Therapy Trial. Heart Rhythm. 2017 Dec;14(12):1820-1825. doi: 10.1016/j.hrthm.2017.08.017. Epub 2017 Sep 9. PMID 28893549
- [Derived] Yamasaki H, Lustgarten D, Cerkvenik J, Birnie D, Gasparini M, Lee KL, Sekiguchi Y, Varma N, Lemke B, Starling RC, Aonuma K. Adaptive CRT in patients with normal AV conduction and left bundle branch block: Does QRS duration matter? Int J Cardiol. 2017 Aug 1;240:297-301. doi: 10.1016/j.ijcard.2017.04.036. Epub 2017 Apr 12. PMID 28416247
- [Derived] Starling RC, Krum H, Bril S, Tsintzos SI, Rogers T, Hudnall JH, Martin DO. Impact of a Novel Adaptive Optimization Algorithm on 30-Day Readmissions: Evidence From the Adaptive CRT Trial. JACC Heart Fail. 2015 Jul;3(7):565-572. doi: 10.1016/j.jchf.2015.03.001. Epub 2015 Jun 10. PMID 26071616
- [Derived] Birnie D, Lemke B, Aonuma K, Krum H, Lee KL, Gasparini M, Starling RC, Milasinovic G, Gorcsan J 3rd, Houmsse M, Abeyratne A, Sambelashvili A, Martin DO. Clinical outcomes with synchronized left ventricular pacing: analysis of the adaptive CRT trial. Heart Rhythm. 2013 Sep;10(9):1368-74. doi: 10.1016/j.hrthm.2013.07.007. Epub 2013 Jul 11. PMID 23851059
- [Derived] Krum H, Lemke B, Birnie D, Lee KL, Aonuma K, Starling RC, Gasparini M, Gorcsan J, Rogers T, Sambelashvili A, Kalmes A, Martin D. A novel algorithm for individualized cardiac resynchronization therapy: rationale and design of the adaptive cardiac resynchronization therapy trial. Am Heart J. 2012 May;163(5):747-752.e1. doi: 10.1016/j.ahj.2012.02.007. PMID 22607850

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number of:
  * 522 pts enrolled, 1 exit
  * 521 pts with baseline information, 16 exits
  * 505 pts of which 14 unsuccessful implants and 491 successful implants, 12 exits and 1 death
  * 478 randomized (318 to aCRT, 160 to control)
Groups:
- Adaptive CRT (aCRT) Pacing: Cardiac resynchronization therapy (CRT) with adaptive pacing
  Cardiac Resynchronization Therapy-Defibrillator (CRT-D): Market approved Medtronic Vision 3D™ CRT-D implantable device (Consulta® CRT-D, Maximo II® CRT-D, or Concerto II® CRT-D)
  Adaptive CRT (aCRT) Pacing: Adaptive CRT pacing software adjusts how the device paces the heart based on the patient's current heart status
- Standard Biventricular Pacing: Cardiac resynchronization therapy (CRT) with biventricular pacing only (without adaptive pacing)
  Cardiac Resynchronization Therapy-Defibrillator (CRT-D): Market approved Medtronic Vision 3D™ CRT-D implantable device (Consulta® CRT-D, Maximo II® CRT-D, or Concerto II® CRT-D)
Period: Overall Study
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
Started | 318 | 160
Completed | 299 | 155
Not Completed | 19 | 5
Not completed — Death | 13 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing | Total
Number analyzed (Participants) | 318 | 160 | 478
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (11.2) | 66.2 (9.7) | 65.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 51 | 148
  Male | 221 | 109 | 330
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 3 | 11
  Black or African American | 29 | 6 | 35
  Hispanic or Latino | 13 | 5 | 18
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  White or Caucasian | 257 | 139 | 396
  Two or more races | 3 | 1 | 4
  Other race | 0 | 0 | 0
  Not available | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  Russia | 1 | 0 | 1
  Hong Kong | 2 | 1 | 3
  United States | 176 | 87 | 263
  Japan | 4 | 2 | 6
  Spain | 1 | 0 | 1
  Saudi Arabia | 1 | 1 | 2
  Canada | 17 | 8 | 25
  Austria | 5 | 2 | 7
  Netherlands | 11 | 5 | 16
  Sweden | 2 | 2 | 4
  Belgium | 6 | 3 | 9
  Norway | 7 | 3 | 10
  Denmark | 11 | 7 | 18
  Italy | 3 | 2 | 5
  Australia | 18 | 12 | 30
  Serbia | 23 | 10 | 33
  Germany | 31 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Improved Heart Failure Outcomes Clinical Composite Score
Description: Patients considered worsened if they died, were hospitalized with worsening heart failure (HF), crossed over to other arm, demonstrated worsening in New York Heart Association (NYHA) functional class, or reported moderately/markedly worse on 'patient global assessment' compared to before CRT implant. Patients are improved if they are not worsened and have an improved NYHA or reported moderately/markedly improved on the 'patient global assessment' compared to before CRT implant
  Global assessment question for the patient: Specifically in reference to your heart failure symptoms, how do you feel today as compared to how you felt before your CRT system was implanted? O Markedly improved O Moderately improved O Mildly improved O No change O Slightly worse O Moderately worse O Markedly worse
Time Frame: randomization to six month visit
Measure: Count of Participants; unit: Participants
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
Number analyzed (Participants) | 318 | 160
Participants | 234 | 114
Statistical Analysis 1: Comparison: Adaptive CRT (aCRT) Pacing vs Standard Biventricular Pacing; Test type: Non-Inferiority — The non-inferiority margin was 12%; p = 0.0002, Farrington-Manning test of two ind. prop

2. Primary Outcome: Correlation Between Aortic Velocity Time Integral (AoVTI) at Adaptive CRT and Echo-optimized Device Settings
Description: Correlation between aortic velocity time integral (AoVTI) at Adaptive CRT and echo-optimized device settings. AoVTI is an echocardiographic representative of stroke volume and cardiac performance.
Time Frame: randomization visit and six month visit
Population: Concordance correlations have been calculated between AoVTI at Adaptive CRT AV and VV settings vs. echo-optimized AV and VV settings at randomization and 6 M. Paired AoVTI measurements were used for concordance correlation analysis, where each subject served as his/her own control. AoVTI was not obtained at both settings for 79 patients.
Measure: Number (95% Confidence Interval); unit: Concordance correlation coefficient
Groups:
- All Randomized Patients: The AoVTI was calculated for each Adaptive CRT subject under two different parameter settings: AV and VV settings determined by Adaptive CRT, and AV and VV settings determined by echo-optimization.
  Subsequently a concordance correlation was calculated and reported, thus this measure cannot be reported per treatment arm.
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 399
Concordance correlation coefficient | 0.93 [0.91 to 0.94]
Statistical Analysis 1: Comparison: All Randomized Patients; Test type: Superiority — The pre-specified minimum objective performance criteria was 0.82; p < 0.0001, t-test, 1 sided

3. Primary Outcome: Percentage of Patients With a Safety Event (Inappropriate AV or VV Delay Settings Related to the aCRT Feature)
Description: For each subject, the Adaptive CRT-determined AV and VV delay settings from randomization up to 183-days post-randomization were evaluated to identify any period of 28-days with a wide delay range (>60 ms)
Time Frame: randomization to 6 months post randomization
Population: 17 participants did not have data available for analysis of this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Adaptive CRT (aCRT) Pacing
Number analyzed (Participants) | 301
Participants | 0

4. Secondary Outcome: Right Ventricular Pacing Percentage
Description: The percentage of time the right ventricle is paced by the device
Time Frame: implant to six months post randomization
Measure: Mean (Standard Deviation); unit: percentage of right ventricle pacing
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
Number analyzed (Participants) | 314 | 160
percentage of right ventricle pacing | 51.3 (37.9) | 95.1 (10.5)
Statistical Analysis 1: Comparison: Adaptive CRT (aCRT) Pacing vs Standard Biventricular Pacing; Test type: Superiority; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Change in Left Ventricular End Systolic Volume Index (LVESVi)
Description: Change in left ventricular end systolic volume index (LVESVi).
Time Frame: baseline to six month visit
Measure: Mean (Standard Deviation); unit: milliliters per meter squared
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
Number analyzed (Participants) | 250 | 123
milliliters per meter squared | -8.3 (23.3) | -10.5 (24.2)
Statistical Analysis 1: Comparison: Adaptive CRT (aCRT) Pacing vs Standard Biventricular Pacing; Test type: Non-Inferiority — The non-inferiority margin is 15; p < 0.0001, t-test, 1 sided

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF)
Time Frame: baseline to six month visit
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
Number analyzed (Participants) | 250 | 123
percent | 3.9 (10.0) | 2.9 (9.8)
Statistical Analysis 1: Comparison: Adaptive CRT (aCRT) Pacing vs Standard Biventricular Pacing; Test type: Non-Inferiority — The non-inferiority margin is 2.5; p = 0.0009, t-test, 1 sided

7. Secondary Outcome: Change in New York Heart Association (NYHA) Classification
Description: The New York Heart Association (NYHA) Functional Classification places patients in one of four categories based on how much they are limited during physical activity.
  Class - Patient Symptoms I - No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II- Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III- Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV- Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: baseline to six month visit
Measure: Mean (Standard Deviation); unit: NYHA class
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
Number analyzed (Participants) | 296 | 153
NYHA class | -1.0 (0.8) | -0.8 (0.8)
Statistical Analysis 1: Comparison: Adaptive CRT (aCRT) Pacing vs Standard Biventricular Pacing; Test type: Non-Inferiority — The non-inferiority margin is 0.3; p < 0.0001, t-test, 1 sided

8. Secondary Outcome: Change in Distance Walked During the Six Minute Hall Walk
Time Frame: baseline to six month visit
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
Number analyzed (Participants) | 284 | 142
meters | 42.4 (103.3) | 29.0 (123.0)
Statistical Analysis 1: Comparison: Adaptive CRT (aCRT) Pacing vs Standard Biventricular Pacing; Test type: Non-Inferiority — The non-inferiority margin is 30; p = 0.0002, t-test, 1 sided

9. Secondary Outcome: Change in Quality of Life Measured by the Minnesota Living With Heart Failure Questionnaire (MLWHF)
Description: The MLWHF is a 21 question survey. Scores range from 0-105, with lower scores indicating better health.
Time Frame: baseline to six month visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
Number analyzed (Participants) | 261 | 135
units on a scale | -19.3 (20.7) | -17.6 (23.8)
Statistical Analysis 1: Comparison: Adaptive CRT (aCRT) Pacing vs Standard Biventricular Pacing; Test type: Non-Inferiority — The non-inferiority margin is 5.1; p = 0.002, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: From randomization to the end of the study, which was 31.3 months for the longest-randomized patient. The average follow-up time was 20.2 months.
Arm/Group | Adaptive CRT (aCRT) Pacing | Standard Biventricular Pacing
All-Cause Mortality (participants affected / at risk) | 35/318 | 19/160
Serious Adverse Events (participants affected / at risk) | 158/318 | 86/160
Other Adverse Events (participants affected / at risk) | 50/318 | 34/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adaptive CRT (aCRT) Pacing (N=318) | Standard Biventricular Pacing (N=160)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 2 (2)
Angina pectoris (Cardiac disorders) | 3 (3) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 5 (8)
Atrial flutter (Cardiac disorders) | 4 (5) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure (Cardiac disorders) | 63 (112) | 35 (58)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 7 (7) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 3 (3)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 8 (8) | 4 (6)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 4 (5)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 6 (6) | 4 (4)
Device capturing issue (General disorders) | 1 (1) | 0 (0)
Device connection issue (General disorders) | 0 (0) | 2 (2)
Device dislocation (General disorders) | 11 (11) | 7 (10)
Device electrical impedance issue (General disorders) | 1 (1) | 0 (0)
Device lead damage (General disorders) | 1 (1) | 1 (1)
Device misuse (General disorders) | 1 (1) | 1 (1)
Device pacing issue (General disorders) | 0 (0) | 1 (1)
Device psychogenic complication (General disorders) | 0 (0) | 1 (1)
Device stimulation issue (General disorders) | 2 (2) | 2 (2)
Hernia (General disorders) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 2 (2) | 1 (1)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Polyp (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) | 1 (1)
Undersensing (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 4 (4)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 16 (19) | 9 (12)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (9) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pocket erosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin abnormal (Investigations) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Cervical root pain (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 6 (7) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 8 (9) | 6 (6)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 6 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Heart transplant (Surgical and medical procedures) | 3 (3) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adaptive CRT (aCRT) Pacing (N=318) | Standard Biventricular Pacing (N=160)
Atrial fibrillation (Cardiac disorders) | 10 (10) | 14 (15)
Cardiac failure (Cardiac disorders) | 28 (33) | 14 (15)
Device stimulation issue (General disorders) | 14 (17) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and Participating Institutions will provide any publication of Study Data generated by PI and/or Participating Institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.